CLINICAL TRIAL: NCT03875352
Title: The Influence of Nursing Technique Applied at the Central Venous Catheter Insertion Site Upon the Incidence of Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KHO-01-CVC; RVO-FNOs/2016 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2019-03-10; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Surgery; Multiorgan Failure; Haematologic Disease
Keywords: central venous catheter; reddening; dressing; hydrophilic methacrylate gel; chlorhexidine gluconate
MeSH Terms: conditions — Multiple Organ Failure; Hematologic Diseases

STUDY DESIGN:
Intervention Model Description: The study subjects were randomized into two study arms, in both of which two interventions were performed.
Masking Description: The study was designed as open-label, no masking was used in the protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neutropenia patients (Experimental): Patients with neutropenia were treated using the CHG and HMG technique.
  Interventions: Procedure: CHG technique; Procedure: HMG technique
- No neutropenia patients (Experimental): Patients with no neutropenia were treated using the CHG and HMG technique.
  Interventions: Procedure: CHG technique; Procedure: HMG technique

INTERVENTIONS:
Procedure: CHG technique — The CHG technique includes treatment using dressing with chlorhexidine.
Procedure: HMG technique — The HMG technique includes treatment using hydrophilic methacrylate gel and transparent foil.

SUMMARY:
Assessing the impact of the nursing technique applied at the insertion site of the central venous catheter using hydrophilic methacrylate gel (HMG) and 2% Chlorhexidine (CHG) upon the incidence of inflammatory complications when treating the surrounding of the central venous catheter.

DETAILED DESCRIPTION:
The study was a prospective and randomized clinical trial. The study was performed at two departments of the University Hospital Ostrava.

The design and performance of the study were approved by the Ethics Committee of the University Hospital Ostrava.

The patients indicated for insertion of central venous catheter (CVC) were informed about the possible nursing techniques applied at the insertion site of the central venous catheter, participation in the study was conditioned with signing a written informed consent. The study evaluated the superiority of a new procedure in providing nursing care for patients with CVC.

Basic patient characteristics were observed and recorded according to the protocol of the study (age, sex, diagnosis), the number of days with CVC inserted, type of dressing, APACHE II score, the presence of neutropenia and the final score of assessment of local signs of inflammation, which was defined as follows:

0 points = No reddening

1. point = Reddening below 2 mm in diameter around the incision
2. points = Reddening below 5 mm in diameter around the incision
3. points = Reddening exceeding 5 mm in diameter around the incision
4. points = Purulent secretion, swelling, pain
5. points = Catheter sepsis The investigators also recorded the day when the first signs of local infection were observed.

The obtained results were evaluated with standard statistical techniques (Chí-quadrate test, Fisher's exact test).

Upon inserting CVC, the type of draping was recorded (small, middle, large), and the cannulated vein (vena subclavia, left and right, vena jugularis interna, left and right, vena femoralis, left and right). A smear was obtained from around the incision site in all patients after insertion and after extraction; the smears were sent for microbiology cultivation and determination of sensitivity to antibiotic therapy. Changing of the dressings was performed in accordance with standard operating procedures of the University Hospital Ostrava. The CVC was attended under aseptic conditions, using sterile material. Surrounding of CVC was mechanically cleaned and disinfected using 2% chlorhexidine for disinfection of the skin, let to dry, and semipermeable foil was placed at the site, containing chlorhexidine gluconate. The dressing was identified with a date when it was applied. This was left in situ for 3-4 days, and the procedure was repeated.

The patients were randomized into two study groups:

1. HMG Group - the patients were treated with 2% chlorhexidine for skin disinfection, HMG and transparent foil
2. CHG Group - the patients were treated with 2% chlorhexidine for skin disinfection and dressing with CHG The randomization procedure further divided the patients into two study arms

1. Neutropenia Group (defined as the number of neutrophil granulocytes below 1x109/l 2. No-neutropenia Group (with a normal number of neutrophil granulocytes

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patients with CVC
* Hospitalization at ICU

Exclusion Criteria:

* Allergy to HMG
* Allergy to transparent foil
* CVC insertion shorter than 3 days
* Strong bleeding from CVC insertion site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Local signs of inflammation | 3 days at minimum, up to 15 days
  The local signs of inflammation were observed in both study arms and both interventions, and were assessed according to the scoring system described in detail description.

CONTACTS AND LOCATIONS:
Overall Officials: Kateřina Hašová, Mgr., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
The investigators have decided not to make individual participant data available to other researchers.

REFERENCES:
- [Background] Chambers ST, Sanders J, Patton WN, Ganly P, Birch M, Crump JA, Spearing RL. Reduction of exit-site infections of tunnelled intravascular catheters among neutropenic patients by sustained-release chlorhexidine dressings: results from a prospective randomized controlled trial. J Hosp Infect. 2005 Sep;61(1):53-61. doi: 10.1016/j.jhin.2005.01.023. PMID 16002181
- [Background] Crawford AG, Fuhr JP Jr, Rao B. Cost-benefit analysis of chlorhexidine gluconate dressing in the prevention of catheter-related bloodstream infections. Infect Control Hosp Epidemiol. 2004 Aug;25(8):668-74. doi: 10.1086/502459. PMID 15357159
- [Background] Ho KM, Litton E. Use of chlorhexidine-impregnated dressing to prevent vascular and epidural catheter colonization and infection: a meta-analysis. J Antimicrob Chemother. 2006 Aug;58(2):281-7. doi: 10.1093/jac/dkl234. Epub 2006 Jun 6. PMID 16757502
- [Background] Lorente L, Henry C, Martin MM, Jimenez A, Mora ML. Central venous catheter-related infection in a prospective and observational study of 2,595 catheters. Crit Care. 2005;9(6):R631-5. doi: 10.1186/cc3824. Epub 2005 Sep 28. PMID 16280064
- [Background] Mermel LA. What is the predominant source of intravascular catheter infections? Clin Infect Dis. 2011 Jan 15;52(2):211-2. doi: 10.1093/cid/ciq108. PMID 21288845